CLINICAL TRIAL: NCT00332111
Title: Infectious Outcomes Following Pancreas Transplantation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 0603103
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Transplantation
Keywords: transplant; pancreas

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed protocol aims to characterize the infectious episodes in pancreas transplant recipients under the current medical care. Knowing these patients infectious risks, the types of infections that commonly affect them and the morbidity and mortality associated with it will provide valuable information in the evaluation of the safety and efficacy of the current practices. The information generated by this study will also serve as the basis for development of strategies targeting prophylaxis of infectious episodes.

DETAILED DESCRIPTION:
The objectives of the study are:

1. To determine what is the frequency of infectious complications following pancreas transplantation
2. Characterize the clinical and microbiological aspects of the infectious complications following pancreas transplantation
3. Identify predictors for infection following pancreas transplantation
4. Determine the frequency of graft loss and associated mortality of infectious complications following pancreas transplantation

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreas with or without kidney transplantation at the University of Pittsburgh Medical Center from January 1st 2002 to December 31st 2005
* Patients must be above 18 years of age
* Patients undergoing retransplantation may be included.

Exclusion Criteria:

* History of pancreas transplantation at another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pancreatic and kidney transplants
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
30 day outcomes after transplantation | 30 days
  outcomes of transplant patients post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States